CLINICAL TRIAL: NCT06053944
Title: Functional Diagnostic Accuracy of Ultrasonic Flow Ratio in Assessment of Left Main Coronary Artery Stenosis
Acronym: FUNCTION II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-12M-C&T-B-043
Record Dates: First submitted 2023-09-17; First posted 2023-09-26 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-09

CONDITIONS: Left Main Coronary Artery Disease
Keywords: intravascular ultrasound; ultrasonic flow ratio; fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: fractional flow reserve (FFR); ultrasonic flow ratio (UFR); intravascular ultrasound (IVUS) — UFR is a novel IVUS-derived modality for fast computation of FFR without pressure wires and adenosine.

SUMMARY:
This is a prospective, observational, single-center study. The main purpose of this study is to evaluate the diagnostic accuracy of offline computational ultrasonic flow ratio (UFR) in predicting functionally significant left main (LM) coronary stenosis with conventional pressure wire-based fractional flow reserve (FFR) as the standard reference. The study will be conducted in Fuwai Hospital, and a total of 120 patients with intermediated left main coronary vessel diameter stenosis ≥30% and ≤80% are planned to be recruited. Participants who meet the inclusion criteria and do not meet the exclusion criteria will undergo intravascular ultrasound (IVUS) followed by FFR examination. IVUS imaging will be sent to an independent core laboratory for UFR calculation. UFR analyses were performed offline in a blinded fashion without awareness of FFR measurement. Using FFR≤0.80 as the gold standard, the sensitivity and specificity of UFR in the functional significance of left main coronary artery stenosis will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris, unstable angina pectoris, or after the acute phase of myocardial infarction
* Age ≥18 years
* Written informed consent
* Intermediated left main coronary lesions (diameter stenosis of 30%-80% by visual estimation from coronary angiography)

Exclusion Criteria:

* Ineligible for diagnostic IVUS or FFR examination
* Prior coronary artery bypass grafting of the interrogated vessels
* Myocardial infarction within 72 h of coronary angiography
* Severe heart failure
* Serum creatinine levels >150 umol/L, or glomerular filtration rates <45 ml/ kg/1.73 m2
* Allergy to the contrast agent or adenosine
* Life expectancy < 2 years
* Proximal LAD diffuse lesions (diameter stenosis > 50%)
* IVUS pullback not covering the entire lesion
* Severe myocardial bridge in the interrogated vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years of age who will be admitted for coronary angiography and had an indication for FFR measurement at the Fuwai Hospital, Beijing, China, due to stable angina or unstable angina will be consecutively enrolled.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of UFR in predicting functionally significant left main coronary stenosis, using FFR as the reference standard | Immediately after the procedure
  Diagnostic accuracy is defined as UFFR (≤0.80 or >0.80) to identify hemodynamically-significant left main coronary stenosis with FFR (≤0.80 or >0.80) as the reference standard.
Sensitivity and specificity of UFR in predicting functionally significant left main coronary stenosis, using FFR as the reference standard | Immediately after the procedure
  Sensitivity is defined as the proportion of UFR ≤ 0.80 in vessels with hemodynamically-significant stenosis as measured by FFR (FFR ≤ 0.80); specificity is defined as the proportion of UFR > 0.80 in vessels without hemodynamically-significant stenosis as measured by FFR (FFR > 0.80).

SECONDARY OUTCOMES:
Comparison of sensitivity and specificity of UFR and IVUS-derived minimal lumen area (MLA) in predicting functionally significant left main coronary stenosis, using FFR as the reference standard | Immediately after the procedure
  Sensitivity is defined as the proportion of UFR ≤ 0.80 in vessels with hemodynamically-significant stenosis as measured by FFR (FFR ≤ 0.80); specificity is defined as the proportion of UFR > 0.80 in vessels without hemodynamically-significant stenosis as measured by FFR (FFR > 0.80).
The AUC of UFR for left main coronary stenosis with FFR as the gold standard | Immediately after the procedure
  AUC is defined as the area under the receiver-operating characteristic curve.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qian, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Select A State, China